CLINICAL TRIAL: NCT06809062
Title: ApoE Genotyping Analysis in Patients with Suspected Non-haemorrhagic Amyloid Angiopathy
Acronym: CAA-WMH-ApoE
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2024/DR-04
Record Dates: First submitted 2025-01-24; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Amyloid Angiopathy
Keywords: Cerebral Amyloid Angiopathy
MeSH Terms: conditions — Amyloid angiopathy; Cerebral Amyloid Angiopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ischaemic microangiopathy: The study is aimed at patients with manifestations related to a vascular accident visible on MRI.

SUMMARY:
Ischaemic microangiopathic features have recently been incorporated into the criteria for cerebral amyloid angiopathy (CAA).

ApoE genotyping (presence of the E4 allele) is routinely used to help determine the aetiology of a haemorrhagic microangiopathy found on MRI.

Chronic ischaemic disease in CAA is characterised by the presence of :

* multispot pattern on the FLAIR sequence
* severe periventricular FLAIR hypersignals with posterior predominance

The main aim of this study was therefore to analyse the frequency of the presence of one (or two) E4 allele(s) on ApoE genotyping in patients with suspected CAA based on ischaemic MRI involvement with a typical radiological pattern.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischaemic stroke (from causes other than CAA, as CAA is not a frequent cause of ischaemic stroke) with associated stigmata of microangiopathy on MRI that may suggest associated CAA.
* Patients treated at Nîmes University Hospital

Exclusion Criteria:

* Patient refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischaemic stroke (from causes other than CAA, as CAA is not a frequent cause of ischaemic stroke) with associated stigmata of microangiopathy on MRI that may suggest associated CAA.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ApoE genotypage | baseline
  To analyse the frequency of the presence of one (or two) E4 allele(s) on ApoE genotyping in patients with suspected AAC. Endpoint: presence of the E4 allele (Yes/No).

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes